CLINICAL TRIAL: NCT04515017
Title: Study on the Value and Mechanism of AS-OCTA in the Evaluation of Filtering Bleb Function and Outcome After Glaucoma Surgery
Brief Title: Evaluation of Filtering Bleb After Glaucoma Surgery by AS-OCTA
Acronym: AS-OCTA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020KYPJ119
Record Dates: First submitted 2020-08-05; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Trabeculectomy
Keywords: Glaucoma; AS-OCTA; TRAB; 5-FU; MMC; Filtering bleb
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
When antihypertensive drugs or laser therapy can not reach the target intraocular pressure, trabeculectomy (TRAB) is still the standard surgical method for glaucoma. The scarring of the operative area is a common reason for the failure of trabeculectomy. After trabeculectomy, maintaining the shape and function of the filtering bleb is an important aspect to maintain the surgical effect. The increase in the number of blood vessels on the filtering bleb and the morphological curvature are often the manifestations of decompensation of the filtering bleb. Angiogenesis in the filtering bleb region plays an important role in surgical incision healing and is related to the accompanying scar formation. Therefore, the evaluation of vascular distribution of filtering blebs is an important index and early parameter to evaluate the success or failure of surgery. With the improvement of detection methods, it is possible to use AS-OCTA to evaluate the function and prognosis of filtering bleb after trabeculectomy. Antimitotic drugs such as 5-fluorouracil (5-FU) or mitomycin C (MMC) have always been the most commonly used clinical drugs, but the side effects caused by their use are not satisfactory. It is still the research direction of glaucoma to find new targets for regulating wound healing and more safe and effective drugs.

DETAILED DESCRIPTION:
Glaucoma is a group of optic nerve diseases characterized by progressive and irreversible degeneration of retinal ganglion cells and their axons. Retinal ganglion cells, RGCs is a kind of central nervous system neuron whose cell bodies are located in the retina and axons make up the optic nerve. When antihypertensive drugs or laser therapy can not reach the target intraocular pressure, trabeculectomy (TRAB) is still the standard surgical method for glaucoma. The scarring of the operative area is a common reason for the failure of trabeculectomy. After trabeculectomy, maintaining the shape and function of the filtering bleb is an important aspect to maintain the surgical effect. The increase in the number of blood vessels on the filtering bleb and the morphological curvature are often the manifestations of decompensation of the filtering bleb. Angiogenesis in the filtering bleb region plays an important role in surgical incision healing and is related to the accompanying scar formation. Therefore, the evaluation of vascular distribution of filtering blebs is an important index and early parameter to evaluate the success or failure of surgery. With the improvement of detection methods, it is possible to use AS-OCTA to evaluate the function and prognosis of filtering bleb after trabeculectomy. Antimitotic drugs such as 5-fluorouracil (5-FU) or mitomycin C (MMC) have always been the most commonly used clinical drugs, but the side effects caused by their use are not satisfactory. It is still the research direction of glaucoma to find new targets for regulating wound healing and more safe and effective drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are over 18 years old and can complete all the tests and examinations.
2. Patients who want to undergo trabeculectomy in accordance with the diagnosis of glaucoma.
3. Intraocular pressure can not be controlled by intraocular pressure lowering drugs and laser therapy (intraocular pressure can not be controlled ≤ 21mmHg).

Exclusion Criteria:

1. Those with a history of ocular trauma, trabeculectomy within 6 months, eye surgery or eye laser within 3 years.
2. The conjunctival state of the proposed surgical area can not support high-quality imaging (signal intensity < 6).
3. Postoperative conjunctival hemorrhage or serious complications, including hyphema, malignant glaucoma, endophthalmitis and so on.
4. The condition of the whole body does not support surgery, such as heart disease, mental illness, malignant tumor, etc.
5. After trabeculectomy, glaucoma drug treatment or reoperation was performed.
6. Pregnant, lactating and pregnant women. Those who refuse to sign the informed consent form or voluntarily withdraw from the study due to discomfort or other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients preparing for trabeculectomy for glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the results of baseline AS-OCTA at different points in time | AS-OCTA was performed before operation, 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks after operation.
  AS-OCTA

SECONDARY OUTCOMES:
Vision | The examination was performed before operation and 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks after operation.
  Changes of visual acuity at baseline and at different time points
Slit lamp microscope | The examination was performed before operation and 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks after operation.
  Changes of baseline slit lamp microscope at different time points
Anterior segment photography | The examination was performed before operation and 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks after operation.
  Photographic changes of anterior segment at baseline and at different time points
Intraocular pressure | The examination was performed before operation and 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks after operation.
  Changes of intraocular pressure at baseline and at different time points
Anterior chamber gonioscope | The examination was performed before operation and 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks after operation.
  Changes of anterior chamber gonioscope at baseline and at different time points
UBM | The examination was performed before operation and 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks after operation.
  UBM changes at baseline and at different time points
fundus color photography | The examination was performed before operation and 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks after operation.
  Changes of fundus color photography at baseline and at different time points
A ultrasound | The examination was performed before operation and 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks after operation.
  Changes of A-ultrasound at baseline and at different times
B ultrasound | The examination was performed before operation and 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks after operation.
  Changes of B-ultrasound at baseline and at different times
visual field | The examination was performed before operation and 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks after operation.
  Changes of visual field at baseline and at different time points

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinreb RN, Khaw PT. Primary open-angle glaucoma. Lancet. 2004 May 22;363(9422):1711-20. doi: 10.1016/S0140-6736(04)16257-0. PMID 15158634
- [Background] Yamazaki M, Omodaka K, Takahashi H, Nakazawa T. Estimated retinal ganglion cell counts for assessing a wide range of glaucoma stages, from preperimetric to advanced. Clin Exp Ophthalmol. 2017 Apr;45(3):310-313. doi: 10.1111/ceo.12852. Epub 2016 Nov 13. No abstract available. PMID 27741375
- See also: Primary open-angle glaucoma — https://pubmed.ncbi.nlm.nih.gov/15158634/
- See also: Estimated retinal ganglion cell counts for assessing a wide range of glaucoma stages, from preperimetric to advanced — https://pubmed.ncbi.nlm.nih.gov/27741375/